CLINICAL TRIAL: NCT06344715
Title: A Phase 1, Multi-center, Open-label, Dose-escalating Study to Evaluate the Safety and Tolerability of Triple Combination Regimen of SL-T10, GX-I7 and Pembrolizumab in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Phase 1 Study Evaluating Safety and Tolerability of SL-T10, GX-I7, and Pembrolizumab Triple Combination in mCRPC.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SL VAXiGEN (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-T10-001_P1
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — efineptakin alfa; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort S1 (Experimental): SL-T10 (3mg, multiple injections, IM), GX-I7 (320 ug 2 injections, IM)
  Interventions: Biological: SL-T10; Biological: GX-I7
- Cohort S2 (Experimental): SL-T10 (6mg, multiple injections, IM), GX-I7 (320 ug 2 injections, IM)
  Interventions: Biological: SL-T10; Biological: GX-I7
- Cohort a' (Experimental): SL-T10 (3mg, multiple injections, IM), GX-I7 (320 ug 2 injections, IM), Pembrolizumab
  Interventions: Biological: SL-T10; Biological: GX-I7; Biological: Pembrolizumab
- Cohort A (Experimental): SL-T10 (6mg, multiple injections, IM), GX-I7 (320 ug 2 injections, IM), Pembrolizumab
  Interventions: Biological: SL-T10; Biological: GX-I7; Biological: Pembrolizumab
- Cohort B (Experimental): SL-T10 (6mg, multiple injections, IM) GX-I7 (720 ug 2 injections, IM) Pembrolizumab
  Interventions: Biological: SL-T10; Biological: GX-I7; Biological: Pembrolizumab
- Cohort C (Experimental): SL-T10 (6mg, multiple injections, IM), GX-I7 (960 ug 2 injections, IM), Pembrolizumab
  Interventions: Biological: SL-T10; Biological: GX-I7; Biological: Pembrolizumab

INTERVENTIONS:
Biological: SL-T10 — A therapeutic DNA vaccine containing three prostate cancer-specific antigen genes and genetic adjuvants
Biological: GX-I7 — A T-cell growth factor
Biological: Pembrolizumab — An immune check point inhibitor
  Arms: Cohort A; Cohort B; Cohort C; Cohort a'

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SL-T10 and GX-I7 or SL-T10, GX-I7 and pembrolizumab in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of SL-T10, GX-I7, and pembrolizumab in combination in patients with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

1. Male patients 19 years of age or older at the date of written informed consent.
2. Patients with histopathologically or cytologically confirmed adenocarcinoma of the prostate, documented by bone or soft tissue lesions.
3. Patients with castration-resistant prostate cancer with a blood testosterone level of less than 50 ng/dL at the screening visit.
4. patients with metastatic castration-resistant prostate cancer (mCRPC) who meet the following criteria (based on PCWG3.0 modified RECIST 1.1)

1) Prior taxane therapy for metastatic prostate cancer or confirmed refusal or inadequacy of such therapy 2) Patients who have received prior docetaxel and at least one of the following agents: abiraterone acetate or enzalutamide before or after docetaxel treatment 3) Patients with progression of prostate cancer during/after prior therapy, in the investigator's judgment, with either of the following, in the internal or external castration state

1. PSA progression defined as at least 2 PSA level increases (≥1 week interval between each test) and a PSA level of ≥2 ng/mL at Screening
2. Advanced soft tissue disease as defined by RECIST 1.1
3. Progressive bone disease defined as ≥2 new lesions on bone scan (per PCWG3)

5. Patients who are on androgen deprivation therapy (ADT) of any kind (patients who have not undergone bilateral orchiectomy must begin internal castration therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists, LHRH antagonists, or anti-androgenic agents, at least 4 weeks prior to Baseline and must continue for the entire duration of the study)

Exclusion Criteria:

1. patient has an active autoimmune disease or is receiving systemic steroid therapy or in immunosuppressive status.
2. Patient has history of chemotherapy, radiation chemotherapy, biological therapy, immunotherapy, or radiation therapy within 4 weeks prior to the screening visit (In case of nitrosoureas or mitomycin, 6 weeks prior to the screening visit)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Baseline to 23 weeks
  Number of participants with treatment-emergent adverse events (TEAEs)
Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0 | Baseline to 48 weeks
  Number of participants with Serious adverse events (SAEs) as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
PSA response rate | Baseline to 48 weeks
  % patients with a reduction in PSA level from baseline by 50% or greater
PSA progression free survival | Baseline to 48 weeks
  The interval from the date of randomisation to the date of first evidence of PSA progression or death from any cause, whichever occurred first.
Radiographic progression free survival | Baseline to 48 weeks
  The interval from the date of disease progression on CT and/or Tc bone scan or death from any cause, whichever occurred first.
Change of induced T-cell responses for SL-T10 vaccine | Baseline to 48 weeks
  Vaccine-induced T-cell responses assessed by immunoassays in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Kwak, MD, phD, Principal Investigator — Seoul National University Hospital; Chang Wook Jeong, MD, phD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No